CLINICAL TRIAL: NCT02439710
Title: Patient Reported Outcomes Burdens and Experiences - Phase 2 - Pilot Feasibility Study
Brief Title: Patient Reported Outcomes Burdens and Experiences - Phase 2
Acronym: PROBE
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: National Hemophilia Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: HIREB-15-260D
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Quality of life measure (survey) — The QoL tool is a questionnaire

SUMMARY:
The Patient Reported Outcomes, Burdens, and Experiences (PROBE) Study aims to develop a new global tool to enhance the direct patient-voice in health care decision-making. Government and private payers increasingly value data based on patient-centered outcomes research as part of the overall cost-benefit evaluation of high-cost care and treatment of diseases such as hemophilia. This emerging dimension of the healthcare environment presents a significant opportunity and urgent need to improve patient organizations' ability to collect and interpret relevant outcomes data. More robust patient reported data will improve advocacy efforts to build comprehensive care programs, promote home treatment and implement preventative treatment regimens thus allowing advocacy arguments to move beyond emotion and anecdote to those grounded in real-world patient experiences and evidence. With the support of the National Hemophilia Foundation, a global team of investigators will lead a patient focused research project to investigate and directly probe patient perspectives on outcomes they deem relevant to their care. Through PROBE, the investigators will develop and seek to validate the reliability, reproducibility and responsiveness of a low cost, easily administrable inventory for collecting patient self-reported outcomes, burdens and experiences in living with hemophilia. The investigators anticipate that the metrics established through PROBE will allow for comparison of patient outcomes within a country over time and cross-sectionally between countries (regionally and globally).

DETAILED DESCRIPTION:
PROBE is the repository of a standardized survey of patients with hemophilia from a group of countries, to be run annually, collecting anonymized information on quality of life measures and treatment modalities. After developing the tool in phase 1 of the project, a pilot feasibility study is hereto described.

Rationale/Goals

Research based on patient-centered data is increasingly valued by government and private payers and utilized in public-policy decisions as part of the cost-benefit justification for high-cost care and treatment. A frequent question of payers is: Will additional investment (to sustain or expand care) improve the lives of persons with hemophilia?

There is a significant need to improve our ability to collect, collate, and interpret relevant patient-centered data to support the implementation of comprehensive care, home treatment and preventative treatment regimens (e.g., prophylaxis). The PROBE study is intended to fill this gap and enhance the direct patient-voice in the delivery of care and move advocacy efforts to sustain and expand care beyond emotion to arguments grounded in evidence and data.

The overall inventory and the specific metrics developed through PROBE will complement the existing global comparative metrics of the World Federation of Hemophilia (WFH) as provided in the WFH Global Survey (e.g., the percent of patients identified vs. expected within a country, amount of treatment products available within a country on a per capita basis, and the ratio of children to adults surviving into adulthood). While the WFH global metrics are valued and useful, they do not provide a complete or direct insight as to how patients are fairing within their health care system. The existing WFH metrics only serve as proxy measures of the impact of care on patient outcomes within a country.

PROBE has an integrated knowledge translation component. This component will be manifested through the development and validation of an inventory able to recode experiential data contributed by patient organizations to a valid foundation for evidence-based decision making (e.g. within Health Technology Assessments [HTAs]). PROBE will also be useful in raising awareness within the community and the public of the impact of treatment for persons living with hemophilia (PWH) and the value of effective prevention.

GENERAL OBJECTIVES OF THE PROBE PROGRAM

The focus of PROBE will be to investigate and directly probe patient perspectives on outcomes they deem relevant to their care. Through PROBE, the investigators will develop and seek to validate the reliability, reproducibility and responsiveness of a low-cost, easily administrable inventory for collecting patient self-reported outcomes, burdens and experiences in living with hemophilia.

A preliminary instrument definition and user testing phase has been completed. This phase has involved an interactive workshop and take-home project utilizing economic concepts and patient reported outcomes (PRO) collection techniques. The workshop was conducted on January 22-23 in Barcelona, Spain. During this workshop, participants partook in an exercise utilizing the PROBE study draft questionnaire developed by the investigators and provided feedback for refinement prior to its finalization for use in the pilot feasibility assessment. During the workshop, the PROBE investigation team sought participant insight on the questionnaire, proposed inventory and study methodology. The workshop also further validated the overall PROBE study goals and better characterized the viability for patient organizations to simply collect self-reported PRO data directly from PWH.

During this exercise, the research protocol was finalized, including inventory, metrics and questionnaire for collection of inventory data. Questionnaire was translated into local languages and explanatory materials to accompany questionnaire was developed.

The questionnaire was developed based on the EQ-5D domains along with an abbreviated set of supplemental questions looking at various demographics, treatment options, and the impacts of hemophilia on a PWH's life.The final questionnaire integrates the EQ-5D-5L with additional domains assessing the impacts of hemophilia on a PWH's life (e.g., pain, independence, educational attainment, employment). The inventory domains, survey instruments, and normative data / comparators selected were identified to reflect those customarily utilized by coverage bodies (e.g. government / private payers, HTAs and Comparative Effectiveness Research). Where feasible, the investigators incorporated generic instruments that are already widely accepted by public policy makers. In developing the questionnaire, the investigators also reviewed available information on questions utilized or published for other research studies and data collection systems (e.g. ATHN, CDC, EHC, EUHASS, HERO, HUGS, WFH).

CURRENT STUDY: PILOT FEASIBILITY STUDY

This is a pilot feasibility study to validate the proof of concept, assess reproducibility and practicality of developing an inventory for large-scale assessment of patient-centered outcomes in PWH. The investigators expect to be able to compare the effect of different treatment delivery modalities and regimens on patient outcomes. The investigators anticipate that the metrics established will allow for comparison of patient outcomes within a country over time and cross-sectionally between countries (regionally and globally), thus providing an important new tool to sustain and promote additional health care investment.

STUDY DESIGN

Twelve countries have been invited to participate i(Australia, New Zealand, France, Hungary, Italy, Spain, The Netherlands, United Kingdom, Argentina, Brazil, Colombia, and Venezuela).

Each participating patient organization has committed to participate in this feasibility project. Six will be selected based on capacity assessment of the local infrastructure.

The final questionnaire will be mailed to each of the participant organization in each of the countries, and administered to 2 groups of 50 subject for each country, three months apart. Questionnaire responses will be returned to a single independent site for analysis, where a central data repository will be established and data analyst retained (McMaster University). Demographic and treatment related information will be collected for correlation analysis and to assess the discriminatory properties of the questionnaire components, but not included in the final tool (inventory).

Two moderate runs of the inventory will be conducted in each country three months apart to demonstrate reproducibility (Approximately 600 PWH in total - 50 PWH per sampling exercise x six countries x two test runs per country). Both paper and web versions will be developed with translations as required. PWH will be recruited for participation via patient organization contact database and their social media portals.

Reproducibility will be assessed based on an analysis of amount of variability within and across sampling exercises with each country. Responsiveness will be assessed based on response rate and percent complete responses. Reliability will be demonstrated by a combined assessment of measurements for the primary outcomes (e.g. response rate, complete responses, agreement between exercises, completion time, cost and feasibility of execution.) (See: Primary Outcome Variables / Measurement Of Results section below).

The data will be collected at the individual level, but responses will be de-identified and aggregated to perform comparison of outcomes at the population level rather than to allow comparison of outcomes at the individual patient level.

Expected results

The PROBE inventory will ideally complement and enhance the utility of the WFH database, providing the opportunity to build a country specific rich data set for comparisons of patient-centered outcomes and provide critical data to support advocacy efforts to improve morbidity, mortality and overall quality of life.

Future applications could include development of a WFH Global Survey style report every 2-3 years providing updated comparative data or a WFH training monograph to support a wider roll-out of the PROBE inventory with National Member Organizations. Additionally, the inventory could be routinely conducted both before commencing and after completion of a country development initiative (e.g. WFH GAP) or implementation of a major health care reform impacting PWH (e.g. introduction of prophylaxis or home treatment) to monitor and compare the impact on patient outcomes.

Once validated, PROBE will establish a mechanism to make the inventory widely available for use within the hemophilia community. However, the specific mechanism to make the PROBE questionnaire and its related methodology available has not yet been established. This may include a system requesting prior consent to use and/or developing a mechanism for collaborative studies.

STUDY POPULATION

Each country will be permitted to determine their target population for the take-home project. The PROBE Investigators will provide guidance on study population parameters, as required. Patients will be recruited according to the final inclusion criteria. No randomization will be required.

There will be approximately 600 PWH in total. The number of PWH participating in each country project will be variable. As this aspect of the PROBE study is an exercise to better understand best practices and obtain learning from execution of patient-centered research in country the number of participants has not been assessed as critical. This number of PWH (600) assumes 12 countries participate in the project.

Moderate / Severe PWH (Age bands or limits may be utilized to narrow the study population). Patients will be recruited according to the final inclusion criteria. No randomization will be required. Two moderate to large test runs of the inventory will be conducted in each country three months apart to demonstrate reproducibility (Approximately 600 PWH in total = 50 PWH per "sampling exercise" x six countries x two test runs per country). PWH participating in each of the two test runs may, but would not necessarily be the same.

When normative data are not available for comparison to the general population, the investigators will consider strategies to produce a comparator (e.g. surveying non-effected siblings). They will also explore suitable data from other chronic conditions to support the aim of the study.

Study results will include an assessment of the adequacy of the small sample size to achieve reproducibility. The study design is intended to describe characteristics generally within the overall study population and not to test for differences in certain attributes of subgroups.

Inclusion Criteria - For both phases, PWH will be recruited through national hemophilia patient organizations utilizing their existing membership rosters, social media outlets and meetings / events. The investigators are not proposing a pre-determined method of PWH recruitment. They will utilize the the information gathered in the workshop and take-home project to inform best practice in recruitment methodology for the next steps of the project. The investigators may consider requesting different countries test different PWH recruitment strategies to test reproducibility.

Exclusion Criteria - Disease severity and Age bands or age limits (e.g. ≥ Age 18) may be utilized to narrow the study population. During the January 2015 meeting of the investigators the inclusion / exclusion criteria will be finalized based on feedback learned during the workshop. Disease severity will be based on patient self-reported severity level.

PRIMARY OUTCOME VARIABLES / MEASUREMENT OF RESULTS

* Response rate (number returned questionnaires/number sent)
* Percent complete responses (number answered question/number answerable questions)
* Time to completion (self-reported completion time, as median and IQR)
* Administrative cost per completed survey (human resources used and dollar-equivalent spent to run the survey)

OTHER STUDY ELEMENTS

* Protected Patient Information - Customary processes will be implemented to protect individual patient identify. No identifiable patient information will be disclosed as part of the study. Data will be collected at the individual PWH level, but responses will be de-identified and aggregated to perform comparison of outcomes at the population level rather than to allow comparison of outcomes at the individual PWH level. Aggregate research results and periodic project updates will be provided to the sponsor. Raw data that could be attributable to individual respondents will not be provided. Independent management and autonomy from sponsor will be assured throughout the project.
* Adverse Event Reporting - Although it is not anticipated that the PROBE Study Team would receive reports of adverse events within the scope of the Study, if the Investigators are made aware of an adverse event involving a product manufactured by a study sponsor through the conduct of the study, the Investigators commit to notify sponsor within one (1) business day of actually becoming aware of any significant product complaint, unexpected adverse event, or governmental investigation or inquiry involving a sponsor's product.
* Institutional Review Board (IRB) Approval - Given the study design only contemplates patients and/or patient organizations directly collecting data from patients and that there is no planned direct Clinician / Hemophilia Treatment Center patient data collection, the investigators do not anticipate the need to require local patient organizations to obtain an IRB approval. They are aware of other global patient-to-patient studies similar to PROBE where IRB approval has not been required.

Two of the primary outcome measures for PROBE are cost and time to completion of the Study. To achieve our goal of developing a low-cost, easily administrable inventory, the investigators will be striving to design a streamlined easily deployable system with minimal up from cost and administrative burdens. PROBE will be mindful that local laws and practices may vary and where required the investigators will comply with local practice for similar type studies. If in the course of PROBE the investigators determine protocols will change sufficiently to require IRB approval the investigators will do so.

FUTURE STEPS

The investigators expect PROBE to be used to perform three comparisons: among countries, within country over time, within country against national normative data. The investigators will preliminarily assess if normative data are available for the domains explored via existing instruments. When normative data are not available, the investigators will consider strategies to produce a comparator (e.g. surveying non-effected siblings). They will also explore suitable data from other chronic conditions to support the aim of the study. They will conduct a sensitivity analysis to assess the sufficiency of the inventory to measure changes on the impact of care within populations of PWH or overtime using data collected from disease specific questions in the PROBE questionnaire in combination with the EQ-5D.

After demonstrating feasibility, a centralized data collection point will be established. Initial data compilation and cleaning of the database will be incorporated within the web-platform development and reporting agreement (e.g. McMaster University). An analyst experienced in analysis of EQ-5D data and the related study domains will conduct an initial analysis. The Investigators will then evaluate the data and determine the final comparisons and correlations for analysis. Supplemental analyses, data correlation and reporting will utilize / be contracted for with a university biostatics or health outcomes department experienced in similar studies (e.g. McMaster University, University of Southern California, North Carolina State University).

Publication plan. The investigators plan to discuss the study results in an end-of-study meeting. A paper will be submitted to Haemophilia summarizing the research findings. Abstracts, posters and requests for oral presentation will be considered for relevant national, regional and international meetings (e.g., EAHAD, EHC, ISPOR, ISTH, NHF, and WFH). They will report the research findings to the participating patient organizations and once validated PROBE will establish a mechanism to make the inventory widely available for use within the hemophilia community.

INVESTIGATION TEAM

A global team of Investigators with diversity of professional and academic credentials* (e.g., quality of life study design, medical, epidemiology, quantitative analysis, legal and health care development) has been assembled.

Principal Investigator:

1. Mark Skinner JD, Institute for Policy Advancement Ltd. (US)

   Co-Investigators:
2. Alfonso Iorio MD Ph.D. FRCPC, McMaster University, Department of Clinical Epidemiology and Biostatistics (Canada)
3. Randall Curtis MBA, Factor VIII Computing (US)
4. Neil Frick MS, National Hemophilia Foundation (US)
5. Michael Nichol Ph.D., University of Southern California, School of Policy and Planning Development (US)
6. Declan Noone, Irish Hemophilia Society (Ireland)
7. David Page, Canadian Hemophilia Society (Canada)
8. Jeff Stonebraker Ph.D., North Carolina State University Poole College of Management (US)
9. Brian O'Mahoney, Irish Hemophilia Society (Ireland)

As noted above, the investigation team includes members with a range of experiences. Specific to designing and testing novel instruments for use in patient outcomes research, the investigators note the following:

* Dr. Nichol (principal investigator) and Mr. Curtis (HUGS Steering Committee co-chair) are associated with the Hemophilia Utilization Group Study (HUGS). A multi-center observational study evaluating the cost of care and burden of illness over the past twenty years. HUGS has developed a number of novel PRO tools. In addition, Dr. Nichol has developed PRO instruments across a range of disorders outside hemophilia.
* Dr. Iorio is a member of the Haemophilia Experiences Results Opportunities (HERO) project which aims to build a comprehensive understanding of life with haemophilia as seen from the perspective of patients, families and caregivers. The HERO questionnaire was novel in its design and implementation via patient organizations.
* Mr. Noone has been a co-investigator and lead author on two multi-national research projects looking at outcomes for patients on prophylaxis, on-demand or combined therapy. Noone et al developed the instrument utilized in the studies.

ELIGIBILITY:
Inclusion Criteria:

* PWH will be recruited through national hemophilia patient organizations utilizing their existing membership rosters, social media outlets and meetings / events. The investigators are not proposing a pre-determined method of PWH recruitment. They will utilize the information acquired in the workshop and take-home project to inform best practice in recruitment methodology for the study. The investigators may consider requesting different countries test different PWH recruitment strategies to test reproducibility.

Exclusion Criteria:

* Disease severity and Age bands or age limits (e.g. ≥ Age 18) may be utilized to narrow the study population. During the January 2015 meeting of the investigators the inclusion / exclusion criteria will be finalized based on feedback learned during the workshop. Disease severity will be based on patient self-reported severity level.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Moderate / Severe PWH (Age bands or limits may be utilized to narrow the study population). Patients will be recruited according to the final inclusion criteria. No randomization will be required. Two moderate to large test runs of the inventory will be conducted in each country three months apart to demonstrate reproducibility. PWH participating in each of the two test runs may, but would not necessarily be the same.
Sampling Method: Non-Probability Sample
Enrollment: 656 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Chai-Adisaksopha C, Skinner MW, Curtis R, Frick N, Nichol MB, Noone D, O'Mahony B, Page D, Stonebraker J, Thabane L, Crowther M, Iorio A. Psychometric properties of the Patient Reported Outcomes, Burdens and Experiences (PROBE) questionnaire. BMJ Open. 2018 Aug 8;8(8):e021900. doi: 10.1136/bmjopen-2018-021900. PMID 30093520
- [Derived] Skinner MW, Chai-Adisaksopha C, Curtis R, Frick N, Nichol M, Noone D, O'Mahony B, Page D, Stonebraker JS, Iorio A. The Patient Reported Outcomes, Burdens and Experiences (PROBE) Project: development and evaluation of a questionnaire assessing patient reported outcomes in people with haemophilia. Pilot Feasibility Stud. 2018 Feb 27;4:58. doi: 10.1186/s40814-018-0253-0. eCollection 2018. PMID 29497561

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through NGOs utilizing their existing membership rosters, social media outlets and meetings or events.
Pre-assignment Details: Participants were required to meet one of two inclusion criteria: (1) PWH (haemophilia A or B with any degree of disease severity) or (2) "Controls" (individuals with no bleeding disorders)
Groups:
- Enrolled Participants: "Patients with hemophilia" (haemophilia A or B with any degree of disease severity) or "Controls" (individuals with no bleeding disorders)
Period: Overall Study
Arm/Group | Enrolled Participants
Started | 656
Completed | 656
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Population: Patients with hemophilia A or hemophilia B with any degree of disease severity or controls
Arm/Group | Enrolled Population
Number analyzed (Participants) | 656
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 646
    Female | 454
    Male | 192
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 35
  Australia | 39
  Brazil | 20
  Canada | 60
  France | 46
  Germany | 17
  Hungary | 34
  Ireland | 38
  Italy | 50
  Japan | 29
  Mexico | 39
  Netherlands | 49
  New Zealand | 43
  Spain | 17
  United Kingdom | 22
  United States | 84
  Venezuela | 34
Years of education [Mean (Standard Deviation); unit: years] | 14.58 (4.67)
Marital status (married) [Count of Participants; unit: Participants] | 421

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: number of filled questionnaires compared to the total number that were sent out
Time Frame: 1 year
Population: patients with hemophilia (hemophilia A or B with any degree of disease severity) or controls
Measure: Count of Units; unit: Questionnaires
Units Other Than Participants: Questionnaires
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 656
Number analyzed (Questionnaires) | 1871
Questionnaires | 656

2. Primary Outcome: Number of Participant Completing the Questionnaire Within 15 Minutes
Description: Number of participants completing the questionnaire within 15 minutes
Time Frame: Up to 15 minutes
Measure: Number; unit: participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 656
participants | 474

3. Primary Outcome: Cost Per Completed Survey
Description: Human and financial resources used by local organization to run the survey - measured as median and full range
Time Frame: 1 year
Measure: Median (Full Range); unit: Dollars (USD) per participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 656
Dollars (USD) per participants | 8.50 [1.20 to 64.30]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Although it is not anticipated that the PROBE Study Team would receive reports of adverse events within the scope of the Study, if the Investigators are made aware of an adverse event involving a product manufactured by a study sponsor , the Investigators commit to notify sponsor within one (1) business day of actually becoming aware of any significant product complaint, unexpected adverse event, or governmental investigation or inquiry involving a sponsor's product.
Arm/Group | Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 0/656
Serious Adverse Events (participants affected / at risk) | 0/656
Other Adverse Events (participants affected / at risk) | 0/656

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT02439710/Prot_SAP_000.pdf